CLINICAL TRIAL: NCT04309357
Title: Evaluation of Thrombolytic Therapy in Acute Ischemic Stroke Outcome: A Cohort Study From North of Iran
Brief Title: Thrombolysis Outcome in Ischemic Stroke
Acronym: TOSSI
Status: Completed | Type: Observational
Sponsor: Mazandaran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Athena Sharifi Razavi, Assistant Professor in neurology, Mazandaran University of Medical Sciences
Other Study IDs: 2464
Record Dates: First submitted 2020-03-12; First posted 2020-03-16 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Stroke, Acute; Thrombolytic Therapy; Alteplase; Mortality
MeSH Terms: conditions — Stroke | interventions — Tissue Plasminogen Activator

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Alteplase — Alteplase in dose 0.9 mg/kg in acute ischemic patient with indications of thrombolytic therapy
  Other Names: recombinant tissue plasminogen activator

SUMMARY:
Consecutive patients with diagnosis of acute ischemic stroke and candidate of thrombolytic therapy during Jan 2017-Mar 2019 in BuAli Sina Hospital ,Sari, Iran, enrolled to this cohort study.

The demographic data, stroke characteristis, lab data and ... recorded. Then patients evaluate every 3 month until 12 month for fallow up.

DETAILED DESCRIPTION:
The variables of the study, including demographic characteristics, risk factors, complete drug history, nosocomial infection and other in-hospital events, hemorrhagic complications, duration of hospitalization,door to needle time, symptom to needle time, clinical and imaging characteristics of resent stroke, laboratory data including fasting blood glucose, lipid profile (total cholesterol, triglyceride, LDL, HDL), hematology markers (CBC diff, HGB, platelet), coagulation markers (PT, PTT, INR), liver function test (ALT, AST, ALP, Bill) and renal function test (BUN, Cr, Cr cl) were collected. All patients underwent a brain computed tomography scan early on the admission and after 24 hours. Cardiological evaluation including Electrocardiogram and echocardiography performed for all patients. Carotid and vertebrobasillar assessed by Doppler ultrasound or magnetic resonance angiography (MRA).

Stroke severity estimated by using modified Rankin Scale (mRS) and National Institutes of Health Stroke Scale(NIHSS) scores on the first day of admission and at discharge by a neurology resident. Then patient evaluate every 3 months until 12 m for fallow up and in each visit vital sign, patient clinical status, any event, Barthel index was recorded.

Safety endpoints of this study were any adverse events clinically relevant to alteplase, specially hemorrhagic complications.

All patients who met all inclusion and exclusion criteria treated with 0.9 mg/kg recombinant tissue plasminogen activator (Actilyse, Boehringer Industry, Germany) up to maximum of 90 mg, 10% of which was injected as a blous dose and remainder infused over an hour.

Primary outcome of this study was alteplase effect in reduce morbidity rate defined by NIHSS and mRS score reduction and rate of functional independence at 3,6 and 12 months Barthel index in fallow up. Minimal clinically important difference defined as reduce NIHSS score at least 25% or MRS score 2 point at discharge day in comparison to admission day. In fallow up evaluations Barthel index 85-100 was considered favorable outcome. Binary outcomes included independence compared with disability or death.

Secondary outcome was rtPA therapy safety that assessed by fatal intra cranial hemorrhage. Also, mortality rate, intracranial hemorrhage rate, any hemorrhagic event rate and any adverse event rate assessed.

ELIGIBILITY:
Inclusion Criteria:

1. writen inform consent
2. diagnosis of acute ischemic stroke by neurologist
3. met all criteria of thrombolytic therapy
4. resived full dose of alteplase

Exclusion Criteria:

1. any contraindication of thrombolytic therapy
2. resived lower than 0.9 mg/kg alteplase

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patient with diagnosis of acute ischemic stroke that met all criteria of thrombolytic therapy, that reffered to Bu Ali Sina hospital during jan 2017-mar 2019, enrolled to this study
Sampling Method: Probability Sample
Enrollment: 214 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Ischemic stroke outcome | 3 months
  evaluation of alteplase effect in morbidity of patient by using barthel index

SECONDARY OUTCOMES:
ischemic stroke mortality | 3 months
  mortality of patients who received alteplase
frequency of adverse event | 3 months
  number of any adverse event of alteplase during study
frequency of fatal adverse event | 3 months
  number of fatal adverse event of alteplase during study

CONTACTS AND LOCATIONS:
Overall Officials: Sharifi-Razavi, Principal Investigator — Mazandaran University of Medical Science
Locations (1):
- Bu Ali Sina hospital , Mazandarn University of Medical Science, Sari, Iran